CLINICAL TRIAL: NCT04974164
Title: Effectiveness of COVID-19 Vaccine (Vero Cell), Inactivated (CoronaVac) for Preventing Symptomatic SARS-CoV-2 Infections and Hospitalizations in the Dominican Republic - Test-Negative Case-Control Study
Brief Title: Effectiveness of COVID-19 Vaccine for Prevention of COVID-19 in the Dominican Republic
Status: Completed | Type: Observational
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Other Study IDs: CoronaVacTND
Record Dates: First submitted 2021-07-22; First posted 2021-07-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All laboratory antibody and RT-PCR tests will be conducted in the central study lab (Laboratorio de Referencia) in the capital city.Antibody testing on the blood sample will be performed to test anti-SARS-CoV-2 IgGantibody,the remaining serum will be stored in -70℃ (or -40℃) freezer；RT-PCR testing on nasopharyngeal swab will be performed to assess the presence of SARS-CoV-2 RNA；SARS-CoV-2 sequencing testing，the remaining swab for PCR testing will be stored in -70oC (or -40oC) freezer for SARS-CoV-2 sequencing testing to assess protection against variants when the test is available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinic cases group: Those with a positive RT-PCR test will be the test-positive cases or clinic cases (approximate N=700)
  Interventions: Biological: Inactivated COVID-19 Vaccine
- Clinic controls group: Those with a negative RT-PCR test will be the test-negative cases or clinic controls (N=700)
  Interventions: Biological: Inactivated COVID-19 Vaccine

INTERVENTIONS:
Biological: Inactivated COVID-19 Vaccine — Each vial contains 0.5 mL (a single dose) and contains 600SU of inactivated SARS-CoV-2 virus antigen
  Other Names: CoronaVac

SUMMARY:
This study is a multisite ,grouped test-negative case-control , phase Ⅳ clinical trial of an inactivated SARS-CoV-2 vaccine (CoronaVac) manufactured by Sinovac Research and Development Co., Ltd.The purpose of this study is to estimate the protective effectiveness of complete vaccination (measured ≥14 days after the second dose) of CoronaVac against symptomatic SARS-COV-2 infections ,COVID-19 hospitalizations and severe cases.

DETAILED DESCRIPTION:
This study is a multisite,grouped test-negative case-control , phase Ⅳ clinical trial in population aged 18 years and older. The experimental vaccine will be manufactured by Sinovac Research and Development Co.,Ltd.The study is planned to be carried out in ten (10) selected hospitals and their catchment communities in five provinces of the Dominican Republic (DR): National District, La Altagracia, Puerto Plata, Santiago, and Santo Domingo from July 1, 2021 to April 30, 2022 . A total of 1400 subjects will be enrolled with 700 estimated clinic cases who are diagnosed as SARS-CoV-2 infection by real-time polymerase chain reaction (RT-PCR); and 700 estimated clinic controls who have a negative RT-PCR test.And subjects will receive two doses of vaccine for primary immunization .

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* Permanent residents of study provinces;
* Able and willing to provide informed consent to participate in the study;
* Able and willing to provide nasopharyngeal swab and venous blood sample;
* Able and willing to complete a questionnaire survey for collecting information on histories of COVID-19 vaccination and disease;
* Considered as suspected cases of SARS-CoV-2 infections by the physicians in the study clinics according to DR national protocol.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from clinic patients in 10 study hospitals in five provinces. Patients who visit the emergency room (ER), fever or respiratory disease clinics to seek diagnosis or health care for severe acute respiratory infection symptoms or signs and are considered as suspected cases of SARS-CoV-2 based in DR national COVID-19 clinical guideline will be invited to participate in the study, and 1400 clinic participants will be enrolled, 140 from each hospital.
Sampling Method: Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Protective effectiveness of complete vaccination of CoronaVac against symptomatic SARS-COV-2 infections | Day 14 after the second dose
  SARS-COV-2 infections confirmed by real-time polymerase chain reaction (RT-PCR) in newly collected nasopharyngeal swab sample among patients visiting the ER in the study hospitals during the study period without a positive RT-PCR test in the preceding 90 days period
Protective effectiveness of complete vaccination of CoronaVac against COVID-19 hospitalizations and severe cases. | Day 14 after the second dose
  Severe disease (including death), defined as a score >5 in terms of WHO clinical progression scale due to SARS-CoV-2 infection

SECONDARY OUTCOMES:
To profile the circulating strains of SARS-CoV-2 in DR | Day 14 after the second dose
  Circulating strains of SARS-CoV-2 in DR

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Perez-Then, Doctor, Principal Investigator — Ministry of Health
Locations (10):
- Dominican Republic (10):
  - Gral Esp Ntra Sra dela Alt, Higuamo, La Altagracia Province
  - Hospital IMG, Salvaleón de Higüey, La Altagracia Province
  - Moscoso Puello Hospital, Bella Vista, Nacional
  - Felix Maria Goico Hospital, Villa Francisca, Nacional
  - Centro Médico Bournigal, Puerto Plata, Puerto Plata
  - Ricardo Limardo, Sosua, Cabarete, Puerto Plata
  - JoséM.Cabral V Báez, Puñal, Santiago Province
  - Clinica Unión Medica del Norte, Santiago de los Caballeros, Santiago Province
  - Marcelino Vélez Santana, Guerra, Santo Domingo Province
  - Fuerza AéreaDr Ramón Lara, Los Alcarrizos, Santo Domingo Province